CLINICAL TRIAL: NCT04720300
Title: Using a Cluster Randomized Controlled Trial to Evaluate a Travel App's Influence on College Student Commuting to Campus
Brief Title: Evaluating a Travel App's Influence on College Student Commuting to Campus
Acronym: CTRAVELAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Atlantic University (Other)
Responsible Party: Principal Investigator, John Renne, Professor, Department of Urban and Regional Planning and Director, Center for Urban and Environmental Solutions, Florida Atlantic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: G-1905-283549; 1588924-3 (Other: FAU IRB)
Record Dates: First submitted 2020-12-06; First posted 2021-01-22 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Health Behavior
Keywords: Students; Transportation; Academic achievement; Behavior
MeSH Terms: conditions — Health Behavior; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MaaS app (Active Comparator): The Mobility-as-a-Service (MaaS) App will be provided to students in the Intervention Group and is intended to facilitate their use of alternative transportation modes such as public transit, ride-hailing, walking, biking, bike share, and e-scooter share to get to campus. The MaaS App will be downloaded to students' smartphones and will provide real-time, multimodal trip planning to students on demand when they open the app. This means, for instance, that a student can plan a trip that includes driving to a train station, taking the train, and then walking from the alighting train station to their final destination. The app will be white label, i.e. it will have a customized look and feel specific to the participating south Florida colleges, and it will have personalization features so that students can tailor the app to their travel patterns. Students in a cluster assigned to the MaaS group will also receive information concerning housing options. Students complete surveys
  Interventions: Other: MaaS app
- No app (Placebo Comparator): Students receive no app, no housing information, students complete surveys.
  Interventions: Other: No app

INTERVENTIONS:
Other: MaaS app — The MaaS App will be downloaded to students' smartphones and will provide real-time, multimodal trip planning to students on demand when they open the app.
  Arms: MaaS app
Other: No app — students receive no app or housing information
  Arms: No app

SUMMARY:
The Cluster Randomized Controlled Trial (cRCT) portion of the study will focus on evaluating the use of information, marketing, and incentives to shape student travel behavior to campus through the three channels identified in Ajzen's (1991) framework.

DETAILED DESCRIPTION:
The investigators will evaluate whether a package of information, marketing, and incentives shifts student travel behavior to campus over one year, and in turn if these shifts in travel behavior result in improved academic performance.

Specific objectives of the cRCT include evaluating whether the intervention results in relatively:

1. Greater utilization of travel modes alternative to single-occupant vehicle travel (transit, biking, walking, bike-sharing, electric scooters, and carpooling)
2. Lower rates of car ownership
3. Superior college performance--higher grade point averages (GPAs)
4. More credit hours completed
5. Higher retention rates

ELIGIBILITY:
Inclusion Criteria:

* Students who live off-campus and attend any of the following three colleges or universities: Florida Atlantic University (FAU), Broward College (BC), or Palm Beach State College (PBSC).
* Students must plan to be at the same institution for the next academic year.

Exclusion Criteria:

* Students live on campus
* Students will leave their current institution within the next academic year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The rate of students using alternative modes increases. | one academic year
  Percentage of trips taken to campus by alternative modes. Will students in the intervention group, subject to information and marketing incentives as delivered through a MaaS app, be more likely to use alternative modes to reach campus?
Number of students who make more frequent use of alternative modes to campus are associated with increased grade point averages. | one academic year
  Number of students who make more frequent use of alternative modes to campus or who do not own vehicles
Number of students who make more frequent use of alternative modes to campus are associated with increases in credit hours earned. | one academic year
  Number of students who make more frequent use of alternative modes to campus or students who do not own vehicles

SECONDARY OUTCOMES:
The rate of students who own vehicles should decrease. | one academic year
  Student car ownership--Will students in the intervention group, subject to information and marketing incentives as delivered through a MaaS app, reduce their level of car reliance?
Number of students who make more frequent use of alternative modes to campus are associated with increases in retention. | one academic year
  Number of students who make more frequent use of alternative modes to campus or who do not own vehicles
Number of students who make more frequent use of alternative modes to campus are associated with increases in degree completion. | one academic year
  Number of studentswho make more frequent use of alternative modes to campus or students or do not own vehicles

OTHER OUTCOMES:
Self-Reported BMI | one academic year
  Number of students reporting BMI within CDC Healthy guidelines increases.
Self-reported general health | one academic year
  Number of students reporting general health as good, very good, or excellent increases

CONTACTS AND LOCATIONS:
Overall Officials: John L Renne, PhD, Principal Investigator — Florida Atlantic University
Locations (1):
- Florida Atlantic University, Boca Raton, Florida, United States

DOCUMENTS (1):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT04720300/Prot_001.pdf